CLINICAL TRIAL: NCT04859621
Title: Phase II Clinical Trial of Vitamin D3 for Reducing Recurrence of Recurrent Lower Urinary Tract Infections: a Multicenter, Randomized, Placebo-controlled Trial
Brief Title: Phase II Clinical Trial of Vitamin D3 for Reducing Recurrence of Recurrent Lower Urinary Tract Infections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-05
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: Vitamin D3; Recurrent lower urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To ensure that the randomized drug treatment period is double-blind, the study drug and placebo control have the same appearance, smell, and taste. Furthermore, the package and label are also adjusted correspondingly to ensure blindness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin D3 4000 IU (Experimental): 4000IU Vitamin D3 Oral Tablet plus standard antibiotic therapy
  Interventions: Drug: Vitamin D3 4000 IU; Other: standard antibiotic therapy
- Vitamin D3 2000 IU (Experimental): 2000IU Vitamin D3 Oral Tablet plus standard antibiotic therapy
  Interventions: Drug: Vitamin D3 2000 IU; Other: standard antibiotic therapy
- Placebo (Placebo Comparator): Placebo Oral Tablet plus standard antibiotic therapy
  Interventions: Drug: Placebo; Other: standard antibiotic therapy

INTERVENTIONS:
Drug: Vitamin D3 4000 IU — Oral administration, 2 tablet per time, qd, oral administration with the first meal, continuous use for 48 weeks
  Arms: Vitamin D3 4000 IU
Drug: Vitamin D3 2000 IU — Oral administration, 1 tablet of each per time, qd, oral administration with the first meal, continuous use for 48 weeks
  Arms: Vitamin D3 2000 IU
Drug: Placebo — Oral administration, 2 tablet per time, qd, oral administration with the first meal, continuous use for 48 weeks
  Arms: Placebo
Other: standard antibiotic therapy — standard antibiotic therapy

SUMMARY:
The aim of this study was to initially evaluate the optimal dose, efficacy, and safety of vitamin D3 for reducing recurrence of recurrent urinary tract infections (rUTIs).

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is a multiple disease that ranks second only to respiratory infections in infectious diseases and is one of the most common infectious diseases among adults. After the first urinary tract infection, the probability of recurrence within half a year and within one year was as high as 24% and 70%, respectively. Urinary tract infection itself has the characteristics of easy recurrence, which is closely related to the abuse of antibiotics, the generation of bacterial resistance, and the decline of local immune function of mucosa.

In the urinary tract, the antibacterial peptide Cathelicidin is mainly located in the proximal tubules of the kidney and the epithelial cells of the renal pelvis and ureter. LL37 is the only antibacterial peptide present in the human body of the Cathelicidin family, which can be regarded as a natural antibiotic produced by the body. Antibacterial peptides have a broad-spectrum antibacterial effect and can exert antibacterial effects against both Gram-positive and Gram-negative bacteria. Vitamin D intake increases the activity of endogenous antimicrobial peptides. Preclinical cell test of Zensun Sci. & Tech. Co., Ltd. confirmed the induction of LL37 in urethral epithelial cells by vitamin D and its broad-spectrum antibacterial effect. Animal experiments also showed the therapeutic effect of LL37 on UTI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years, including 18 and 75 years;
2. at least 3 episodes of lower urinary tract infection in the last 12 months or at least 2 episodes of lower urinary tract infection in the last 6 months;
3. The symptoms of the latest recurrence of lower urinary tract infection have disappeared after treatment, and the treatment dosage of antibiotics has been stopped, and at least one of the following two conditions has been met:A) The middle urinary bacterial culture is less than 10^5 CFU/mL (accept the examination results after the last improvement);B) Urine white blood cell count is less than 5 /HP, and if it can be measured in routine urine examination, it should be less than 25 /μL;
4. Signed written informed consent;
5. Be able to follow the research protocol.

Exclusion Criteria:

1. Complicated with cardio-cerebrovascular and hematopoietic system and other serious primary diseases;
2. Poor glycemic control (HbA1c >7.5%) with diabetes;
3. Patients with genital tract malformation or acute genital tract infection and genital tract tumor;
4. Patients with urinary system tuberculosis and acute pyelonephritis;
5. Patients with cysto-ureteral reflux or urethral reflux;
6. Patients with polycystic kidney disease, neurogenic bladder, indwelling urethral catheterization, urinary tract stones, tumors or fibrous degeneration, etc., determined by the investigator as urinary tract obstruction;
7. Glomerular filtration rate (MDRD formula).20 mL/min/1.73m2, dialysis or kidney transplantation patients;
8. Chronic liver disease may have potential influence on liver function (bilirubin >;1.5 times upper limit of normal value, aspartate aminotransferase or alanine aminotransferase >2 times the upper limit of normal);
9. Patients with vitamin D3 contraindications, such as hypercalcemia, hypervitaminism, hyperphosphatemia with renal rickets, etc.;
10. Patients with diseases that affect the absorption of vitamin D3 in the small intestine, such as Crohn's disease;
11. receiving immunosuppressive agents or GT;10 mg/d glucocorticoids;
12. had received any other investigational drug therapy or participated in another interventional clinical trial within 30 days prior to screening;
13. Have a history of alcohol or drug abuse or suffer from mental illness;
14. Women of child-bearing age who have planned to become pregnant within 2 years (women of child-bearing age are defined as all women with physical ability to become pregnant), or women who are pregnant or lactating;
15. Circumstances in which subjects are judged by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
UTI recurrent incidence in 48 weeks | 48 weeks
  UTI episodes during 48-week treatment for each subject

SECONDARY OUTCOMES:
Recurrence rate of UTI in 48 weeks | 48 weeks
  Comparing the recurrence rate of UTI between different treatment groups
UTI-free duration in 48 weeks | 48 weeks
  Comparing the number of days from the beginning of the study to the first recurrence of UTI, and the number of days from each recurrence to the next recurrence between different treatment groups.
Cumulative relapse-free ratio | 48 weeks
  Ratio of the cumulative duration of UTI-free period to treatment duration

OTHER OUTCOMES:
Antibiotic treatment during the recurrence of UTI | 48 weeks
  Subjects will be given antibiotics during the recurrence of UTI, type/name and the duration of antibiotic treatment will be compared between different treatment groups.
Symptom score of each episode of recurrent lower urinary tract infection | 48 weeks
  Symptom score of each episode of UTI will be evaluated using an overall impression scale with 7 severity levels ( "a" means the best outcome and "g" as the worst outcome.)
Urinary culture bacterial count | 48 weeks
  Urinary culture bacterial count at each recurrence of UTI
Blood and urine levels of antimicrobial peptides | 48 weeks
  Blood and urine levels of antimicrobial peptides at planned and additional visits

CONTACTS AND LOCATIONS:
Overall Officials: Xian He, MD, Principal Investigator — Zhejiang Provincial People's Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality
  - The Fifth People's Hospital, Shanghai, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine，Chongming Branch, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang